CLINICAL TRIAL: NCT07364227
Title: Comparison of Anterior, Posterior, and Combined Intra-Articular Injection Techniques in Patients With Adhesive Capsulitis
Brief Title: Anterior vs Posterior vs Combined Intra-Articular Injections for Adhesive Capsulitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aslinur Keles Ercisli, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Aslinur Keles Ercisli, MD, PhD, Principal investigator, Fatih Sultan Mehmet Training and Research Hospital
Organization: Fatih Sultan Mehmet Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADC2025
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Adhesive Capsulitis of the Shoulder; Intra Articular Injection
Keywords: Adhesive Capsulitis of the Shoulder; Intra-articular Injection; Frozen Shoulder; Ultrasound; Shoulder Pain
MeSH Terms: conditions — Bursitis; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, controlled, parallel-group clinical trial with three intervention arms. Thirty patients with adhesive capsulitis will be randomly assigned in equal numbers (1:1:1) to receive an intra-articular corticosteroid injection via the posterior approach, the anterior approach, or a combined anterior-posterior approach. Each participant will receive only one type of injection, and outcomes will be assessed at baseline, immediately post-injection, and at weeks 3, 6, and 12.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Posterior Injection (Experimental): Single intra-articular injection with corticosteroid + lidocaine + saline via the posterior glenohumeral approach.
  Interventions: Drug: Intervention Name: Posterior Intra-articular Injection
- Arm B - Anterior Injection (Experimental): Same injection solution administered via the anterior (rotator interval) approach.
  Interventions: Drug: Anterior Intra-articular Injection
- Arm C - Combined Anterior + Posterior Injection (Experimental): Same injection solution administered using both anterior and posterior approaches.
  Interventions: Drug: Combined Anterior + Posterior Intra-articular Injection

INTERVENTIONS:
Drug: Intervention Name: Posterior Intra-articular Injection — A single intra-articular injection consisting of 1 cc corticosteroid, 4 cc 2% lidocaine, and 5 cc saline (total 10 cc) administered via the posterior glenohumeral approach.
  Other Names: Posterior Intra-articular Injection
  Arms: Arm A: Posterior Injection
Drug: Anterior Intra-articular Injection — A single intra-articular injection consisting of 1 cc corticosteroid, 4 cc 2% lidocaine, and 5 cc saline (total 10 cc) administered via the anterior (rotator interval) approach.
  Other Names: Anterior hydrodilatation
  Arms: Arm B - Anterior Injection
Drug: Combined Anterior + Posterior Intra-articular Injection — A single intra-articular injection consisting of 1 cc corticosteroid, 4 cc 2% lidocaine, and 5 cc saline (total 10 cc) administered using both anterior and posterior approaches during the same procedure.
  Other Names: combined joint injection
  Arms: Arm C - Combined Anterior + Posterior Injection

SUMMARY:
This randomized controlled clinical trial aims to compare the efficacy of three different intra-articular injection approaches (anterior, posterior, and combined anterior-posterior) in patients with adhesive capsulitis of the shoulder. Thirty participants will be randomly assigned to one of three groups and treated with a standardized injection solution consisting of corticosteroid, lidocaine, and saline. Clinical outcomes will be evaluated using pain scores, functional scales, and imaging parameters.

DETAILED DESCRIPTION:
Adhesive capsulitis (frozen shoulder) is a disabling condition characterized by progressive pain and stiffness of the glenohumeral joint. Intra-articular corticosteroid injections are frequently used to reduce pain and improve mobility; however, the optimal injection approach remains controversial.

This single-center randomized controlled trial will investigate three different approaches: posterior, anterior, and combined anterior-posterior injections. The primary endpoint is improvement in active and passive range of motion. Secondary endpoints include pain scores (VAS), functional outcome measures (SPADI, qDASH, ASES, Constant-Murley, Scratch Test, Subjective Shoulder Value), and ultrasound evaluation of axillary capsule thickness. Assessments will be performed at baseline, immediately after injection, and at weeks 3, 6, and 12.

ELIGIBILITY:
Inclusion Criteria Age 18-70 years Unilateral shoulder pain and stiffness (symptom duration 1-9 months) NRS pain score ≥ 7/10 Passive range of motion limitation >50% in at least two planes, or >30° restriction in ≥2 planes "Freezing stage" (stage 2 adhesive capsulitis) No analgesic use (NSAIDs, opioids, acetaminophen) within 12 hours before intervention Radiography and/or MRI excluding other pathologies (rotator cuff tear, labral lesion, osteoarthritis, etc.) Exclusion Criteria Secondary adhesive capsulitis (trauma, surgery, systemic disease) Prior shoulder surgery or intra-articular steroid injection within 3 months Bilateral frozen shoulder Neurological disorders (Parkinson's disease, ALS, neuropathies) Malignancy, infection, cellulitis, septic arthritis, acute fracture Cognitive impairment, psychiatric disorders, pregnancy Steroid or local anesthetic allergy Poor glycemic control or other contraindications to steroid injections

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Shoulder Range of Motion (ROM) | Baseline, immediately post-injection, week 3, week 6, week 12
  Change in active and passive shoulder joint range of motion (flexion, extension, abduction, external rotation, internal rotation) measured with a goniometer.

SECONDARY OUTCOMES:
Change in Pain Intensity (NRS) | Baseline, immediately post-injection, week 3, week 6, week 12
  Number Rating Scale (0-10) for pain at rest, during activity, and at night.
Subjective Shoulder Value (SSV) | Baseline, immediately post-injection, week 3, week 6, week 12
  Patient's self-reported percentage of normal shoulder function (0-100%).
Shoulder Pain and Disability Index (SPADI) | Baseline, week 3, week 6, week 12
  Questionnaire assessing pain and disability (0-100 score, higher scores = worse function).
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) | Baseline, week 3, week 6, week 12
  Questionnaire measuring upper limb disability and symptoms (0-100 score, higher = worse).
American Shoulder and Elbow Surgeons (ASES) Score | Baseline, week 3, week 6, week 12
  Composite score including pain and function (0-100, higher = better).
Constant-Murley Shoulder Score | Baseline, week 3, week 6, week 12
  Clinical score combining pain, activities of daily living, strength, and ROM (0-100).
Scratch Test Score | Baseline, immediately post-injection, week 3, week 6, week 12
  Functional test measuring the patient's ability to reach behind the back.
Axillary Capsule Thickness (Ultrasound) | Baseline, immediately post-injection (only).
  Ultrasound measurement of axillary recess capsule thickness on the affected shoulder.

CONTACTS AND LOCATIONS:
Overall Officials: Aslinur keles, MD., PhD, Principal Investigator — Health Sciences University Fatih Sultan Mehmet Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No